CLINICAL TRIAL: NCT02373085
Title: Effect of Systematic Search and Antimicrobial Treatment of Asymptomatic Bacteriuria in Kidney Transplant Recipients in the Incidence of Acute Pyelonephritis: a Pragmatic Prospective Randomized Controlled Study.
Brief Title: Prospective Comparative Study About Treatment of Asymptomatic Bacteriuria in Kidney Transplant Recipients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: López-Medrano, Francisco, M.D. (Individual)
Responsible Party: Principal Investigator, Francisco López Medrano, Lopez-MedranoF, López-Medrano, Francisco, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ABTxR-H12O
Record Dates: First submitted 2015-02-13; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Asymptomatic Bacteriuria
Keywords: Asymptomatic Bacteriuria; Kidney transplant recipients; Pyelonephritis
MeSH Terms: conditions — Pyelonephritis | interventions — Anti-Infective Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Antibiotic adjusted to antibiogram (Experimental): A course of 3-14 days of antimicrobial treatment, according to the antibiogram results, will be prescribed for every episode of asymptomatic bacteriuria beyond 2 months after transplantation and during the first 2 years after transplantation
  Interventions: Other: Antibiotic adjusted to antibiogram
- B: no treatment (No Intervention): No treatment of any episode of asymptomatic bacteriuria beyond 2 months after transplantation in kidney transplant recipients.

INTERVENTIONS:
Other: Antibiotic adjusted to antibiogram — A course of 3-14 days of antimicrobial treatment, according to the antibiogram results, will be prescribed for every episode of asymptomatic bacteriuria during the first 2 years after transplantation.
  Other Names: Anti-infective agents
  Arms: A: Antibiotic adjusted to antibiogram

SUMMARY:
Antimicrobial treatment of asymptomatic bacteriuria (AB) in kidney transplant recipients (KTR) is controversial. The investigators performed a comparative, parallel-group, randomized, open-label study to assess, in a real clinical setting, the feasibility of and benefit derived from systematic search and antimicrobial treatment of all episodes of AB.

DETAILED DESCRIPTION:
All patients undergoing KT between January 2011 and December 2013 in a tertiary-care center with an active transplantation program were systematically searched for AB within the first 2 years after transplantation on a regular basis. During the first 2 months after transplantation all episodes of AB were treated. Thereafter, patients were assigned, according to a computer-generated randomization sequence, to group A (systematic antimicrobial treatment of all episodes of AB) or group B (no treatment). Treatment was chosen according to the results of the urine culture.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients developing asymptomatic bacteriuria beyond 2 months after transplantation.

Exclusion Criteria:

* <18 years old
* Pregnant women
* Kidney-pancreas transplantation
* Double J stent catheterization at the momento of randomization
* Permanent vesical catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Pyelonephritis | 2 years after transplantation
  The number of patients that develope pyelonephritis in the first 2 years after transplantation in each group, divided by the number of patients allocated in each group at randomization.

SECONDARY OUTCOMES:
Incidence of lower tract urinary infection | 2 years after transplantation
  The number of patients that develope lower tract urinary infection in the first 2 years after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of Clostridium difficile infection | 2 years after transplantation
  The number of patients that develope Clostridium difficile infection in the first 2 years after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of multidrug resistant bacteria colonization/infection | 2 years after transplantation
  The number of patients that develope multidrug resistant bacteria colonization/infection in the first 2 years after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Long-term graft function | At 1 year and 2 years after transplantation
  Long-term graft function measured by average serum creatinine at several points until the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco López-Medrano, MD,PhD, Principal Investigator — López-Medrano, Francisco, M.D.

REFERENCES:
- [Derived] Origuen J, Lopez-Medrano F, Fernandez-Ruiz M, Polanco N, Gutierrez E, Gonzalez E, Merida E, Ruiz-Merlo T, Morales-Cartagena A, Perez-Jacoiste Asin MA, Garcia-Reyne A, San Juan R, Orellana MA, Andres A, Aguado JM. Should Asymptomatic Bacteriuria Be Systematically Treated in Kidney Transplant Recipients? Results From a Randomized Controlled Trial. Am J Transplant. 2016 Oct;16(10):2943-2953. doi: 10.1111/ajt.13829. Epub 2016 May 23. PMID 27088545